CLINICAL TRIAL: NCT05721144
Title: Inhaled NO ReDuce postoperatIve pulmoNAry complicATions in patiEnts With Recent COVID-19 Infection
Brief Title: Inhaled NO in Surgical Patients With Recent COVID-19 Infection
Acronym: INORDINATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Principal Investigator, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY-20230079
Record Dates: First submitted 2023-02-07; First posted 2023-02-09 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Nitric Oxide; COVID-19; Surgery; Postoperative Complications
Keywords: Nitric Oxide Inhalation; Postoperative Pulmonary Complications; Surgery; COVID-19
MeSH Terms: conditions — COVID-19; Postoperative Complications | interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Treatment Group (Experimental): Inspired NO/N2 will be delivered at 80 parts per million (ppm) after anesthesia induction and intubation and lasted until the end of surgery and leave the operating room. The physician will follow their own institutional weaning protocols.
  Interventions: Drug: Nitric Oxide Gas
- Sham Comparator: Control Group (No Intervention): The delivery system will be set up anyway without studying gas administration

INTERVENTIONS:
Drug: Nitric Oxide Gas — Inspired NO/N2 will be delivered at 80 parts per million (ppm) after anesthesia induction and intubation and lasted until the end of surgery and leave the operating room.
  Other Names: Nitric Oxide inhalation
  Arms: Experimental: Treatment Group

SUMMARY:
The aim of this study is to evaluate the effect of perioperative inhalation of NO on reducing the incidence of postoperative pulmonary complications in patients with recent COVID-19 infection, and to evaluate whether inhaled NO can improve the prognosis of patients.

The investigators will enroll 660 surgical patients who was infected with SARS-CoV-2 within 42days (7 weeks ) prior to planed surgery under general anesthesia. Patients will be randomized to receive either inhaled nitric oxide (per protocol) or a placebo. Perioperative standards of care will be the institution's own protocols (such as ventilation strategies and use and dose of anesthetics, analgesia and fluid management, etc).

DETAILED DESCRIPTION:
The outbreak of COVID-19 and its global pandemic has posed a threat to public health. On December 7, 2022, the National Health Commission (NHC) of China issued an announcement on further optimization of public health control measures. Since then, the rapid spread and breakthrough of SARS-CoV-2 infections have been observed in the majority of China, caused by the more infectious and less virulent Omicron variant of SARS-Cov-2. Consequently, the proportion of surgical patients with current or previous SARS-CoV-2 infections will inevitably increase within a relatively narrow time window.

It has been reported that a history of SARS-CoV-2 infection is associated with a transiently elevated risk of postoperative complications. The longer the time interval between infection and surgery, the lower the risk of postoperative complications. An updated recommendation suggested postponing surgery for at least seven weeks following SARS-CoV-2 infection, thereby reducing the risk of postoperative complications and 30-day mortality to baseline levels (similar to those without a history of SARS-CoV-2 infection).

COVID-19 infection significantly affects respiratory functions by massively disrupting pulmonary oxygenation and activating the synthesis of proinflammatory cytokines, inducing severe oxidative stress, enhanced vascular permeability, and endothelial dysfunction which has rendered researchers and clinicians to depend on prophylactic treatment due to the unavailability of proper disease management approaches. Inhaled nitric oxide gas (NO) has shown antiviral activity against Coronavirus during the 2003 SARS outbreak. Previous studies have indicated that nitric oxide (NO) application appears to be significant concerning the antiviral activities, antioxidant, and anti-inflammatory properties in relieving disease-related symptoms. Inhaled nitric oxide had been widely used during the Covid-19 pandemic. In the scoping and systemic reviews, it was demonstrated that nitric oxide inhalation was effective in improving oxygenation, cardiopulmonary function, and fastening virus clearance. The investigators designed this study to assess whether inhaled NO reduces postoperative pulmonary complications in patients with a COVID-19 infection history 7 weeks prior to surgery.

Here, the investigators propose a randomized clinical trial aimed to improve postoperative outcomes in patients with an increased risk of postoperative pulmonary complications after COVID-19 infection.

Control group: the institutional standard of care will be delivered. Treatment group: In addition to standard therapy, the subjects will receive inhalation of NO. Inspired NO/N2 will be delivered at 80 parts per million (ppm) after anesthesia induction and intubation and last until the end of surgery and leave the operating room. The physician will follow their own institutional weaning protocols. In the absence of institutional protocols, NO will be reduced in a step-wise fashion starting from 40 ppm to 20, 10, 5, 3, 2, and 1 ppm. If hypoxemia (SpO2 < 93%) or acute hypotension (systolic blood pressure < 90 mmHg) occurs during weaning, NO should be increased to a prior higher concentration.

Safety: prolonged treatment with inhaled NO can lead to increased methemoglobin levels. Blood levels of methemoglobin will be monitored via a non-invasive CO-oximeter or MetHb levels in the blood. If methemoglobin levels rise above 5% at any point in the study, inhaled NO concentration will be halved.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. Planned for surgery under general anesthesia
3. With a history of COVID-19 infection within 7 weeks prior to surgery.

Exclusion Criteria:

1. Physician makes a decision that trial involvement is not in the patient's best interest or any condition that does not allow the protocol to be followed safely
2. ASA ≥ IV, life expectancy< 24 h.
3. Pregnant or lactating women.
4. Severe liver disease (Child-Pugh score ≥ 12).
5. Patients with severe respiratory failure need mechanical ventilation support or ECMO life support before the operation.
6. Severe renal dysfunction (eGFRC≤30 ml/min/1.73m2) or receiving continuous renal replacement therapy, hemodialysis, and peritoneal dialysis.
7. Having received or participated in other clinical trials within the previous month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
postoperative pulmonary complications | within 7 days after operation
  It is composite outcome including respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, and aspiration pneumonitis

SECONDARY OUTCOMES:
mortality within 30 days postoperatively | within 30 days after operation
  All-cause mortality
Classification of pulmonary complications (Clavien-Dindo) | within 7 days after operation
  Evaluation of the severity of pulmonary complications according to Clavien-Dindo classification. It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V).
the rate of unplanned ICU admission | within 7 days after operation
  Percentage of patients admitted into ICU after surgery, which is not expected before surgery
postoperative length of hospital stay | From the date of surgery until the date patient discharge from hospital, assessed up to 30 days
  duration between end of surgery and discharge from hospital
Incidence of thrombotic events | From the date of surgery until the date patient discharge from hospital, assessed up to 30 days
  including DVT and pulmonary embolism
incidence of nonpulmonary complications | From the date of surgery until the date patient discharge from hospital, assessed up to 30 days
  including acute kidney injury, Stroke and myocardial infarction
postoperative comprehensive complication index (CCI) | within 7 days after operation
  Ranging from 0 (no complication) to 100 (death) was computed based on the Clavien-Dindo classification

OTHER OUTCOMES:
Incidence of hypotension | From anesthesia induction until leave operation room, assessed up to 12 hrs
  It is diagnosed as SBP < 90mmHg or drop ≥ 30% of baseline lasted for 5 min
Incidence of hypertension | During surgery, from anesthesia induction to end of anesthesia
  It is diagnosed as SBP > 180 mmHg or rise ≥ 30% of baseline lasted for 5 min
Occurrence of arrhythmia | From anesthesia induction until leave operation room, assessed up to 12 hrs
  consisted of bradycardia (HR < 40bpm) or tachycardia (HR> 100 bpm) or new onset of arrhythmia that require Anti-arrhythmic drugs
Incidence of airway hyperresponsiveness | From anesthesia induction until leave operation room, assessed up to 12 hrs
  airway peak pressure > 40 cm water
Number that the concentration of NO was adjusted | During NO inhalation, from anesthesia induction until leave operation room, assessed up to 12 hrs
  For safety, if the N2O or metHb level exceed safety threshold, the NO concentration needs to be adjusted. The number of adjustment is recorded
massive bleeding | From anesthesia induction until leave operation room, assessed up to 12 hrs
  bleeding exceed 1000 ml

CONTACTS AND LOCATIONS:
Overall Officials: Chong Lei, MD&phD, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in this article, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 12 months
Access Criteria: Investigators who provide a methodologically sound proposal and whose proposed use of data has been approved by the steering of INORDINATE identified for individual participant data meta-analysis. Proposals should be directed to corresponding author of the publication. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Chen L, Liu P, Gao H, Sun B, Chao D, Wang F, Zhu Y, Hedenstierna G, Wang CG. Inhalation of nitric oxide in the treatment of severe acute respiratory syndrome: a rescue trial in Beijing. Clin Infect Dis. 2004 Nov 15;39(10):1531-5. doi: 10.1086/425357. Epub 2004 Oct 22. PMID 15546092
- [Background] Keyaerts E, Vijgen L, Chen L, Maes P, Hedenstierna G, Van Ranst M. Inhibition of SARS-coronavirus infection in vitro by S-nitroso-N-acetylpenicillamine, a nitric oxide donor compound. Int J Infect Dis. 2004 Jul;8(4):223-6. doi: 10.1016/j.ijid.2004.04.012. PMID 15234326
- [Background] Valsecchi C, Winterton D, Safaee Fakhr B, Collier AY, Nozari A, Ortoleva J, Mukerji S, Gibson LE, Carroll RW, Shaefi S, Pinciroli R, La Vita C, Ackman JB, Hohmann E, Arora P, Barth WH Jr, Kaimal A, Ichinose F, Berra L; DELiverly oF iNO (DELFiNO) Network Collaborators. High-Dose Inhaled Nitric Oxide for the Treatment of Spontaneously Breathing Pregnant Patients With Severe Coronavirus Disease 2019 (COVID-19) Pneumonia. Obstet Gynecol. 2022 Aug 1;140(2):195-203. doi: 10.1097/AOG.0000000000004847. Epub 2022 Jul 6. PMID 35852269
- [Background] Fang W, Jiang J, Su L, Shu T, Liu H, Lai S, Ghiladi RA, Wang J. The role of NO in COVID-19 and potential therapeutic strategies. Free Radic Biol Med. 2021 Feb 1;163:153-162. doi: 10.1016/j.freeradbiomed.2020.12.008. Epub 2020 Dec 22. PMID 33347987
- [Background] Al Sulaiman K, Korayem GB, Altebainawi AF, Al Harbi S, Alissa A, Alharthi A, Kensara R, Alfahed A, Vishwakarma R, Al Haji H, Almohaimid N, Al Zumai O, Alrubayan F, Asiri A, Alkahtani N, Alolayan A, Alsohimi S, Melibari N, Almagthali A, Aljahdali S, Alenazi AA, Alsaeedi AS, Al Ghamdi G, Al Faris O, Alqahtani J, Al Qahtani J, Alshammari KA, Alshammari KI, Aljuhani O. Evaluation of inhaled nitric oxide (iNO) treatment for moderate-to-severe ARDS in critically ill patients with COVID-19: a multicenter cohort study. Crit Care. 2022 Oct 3;26(1):304. doi: 10.1186/s13054-022-04158-y. PMID 36192801
- [Background] Garfield B, McFadyen C, Briar C, Bleakley C, Vlachou A, Baldwin M, Lees N, Price S, Ledot S, McCabe C, Wort SJ, Patel BV, Price LC. Potential for personalised application of inhaled nitric oxide in COVID-19 pneumonia. Br J Anaesth. 2021 Feb;126(2):e72-e75. doi: 10.1016/j.bja.2020.11.006. Epub 2020 Nov 14. No abstract available. PMID 33288208
- [Background] Ghosh A, Joseph B, Anil S. Nitric Oxide in the Management of Respiratory Consequences in COVID-19: A Scoping Review of a Different Treatment Approach. Cureus. 2022 Apr 5;14(4):e23852. doi: 10.7759/cureus.23852. eCollection 2022 Apr. PMID 35530860
- [Background] Bunch CM, Moore EE, Moore HB, Neal MD, Thomas AV, Zackariya N, Zhao J, Zackariya S, Brenner TJ, Berquist M, Buckner H, Wiarda G, Fulkerson D, Huff W, Kwaan HC, Lankowicz G, Laubscher GJ, Lourens PJ, Pretorius E, Kotze MJ, Moolla MS, Sithole S, Maponga TG, Kell DB, Fox MD, Gillespie L, Khan RZ, Mamczak CN, March R, Macias R, Bull BS, Walsh MM. Immuno-Thrombotic Complications of COVID-19: Implications for Timing of Surgery and Anticoagulation. Front Surg. 2022 May 4;9:889999. doi: 10.3389/fsurg.2022.889999. eCollection 2022. PMID 35599794
- [Background] COVIDSurg Collaborative; GlobalSurg Collaborative. SARS-CoV-2 infection and venous thromboembolism after surgery: an international prospective cohort study. Anaesthesia. 2022 Jan;77(1):28-39. doi: 10.1111/anae.15563. Epub 2021 Aug 24. PMID 34428858
- [Background] COVIDSurg Collaborative. Outcomes and Their State-level Variation in Patients Undergoing Surgery With Perioperative SARS-CoV-2 Infection in the USA: A Prospective Multicenter Study. Ann Surg. 2022 Feb 1;275(2):247-251. doi: 10.1097/SLA.0000000000005310. PMID 34793350
- [Background] Abbott TEF, Fowler AJ, Dobbs TD, Gibson J, Shahid T, Dias P, Akbari A, Whitaker IS, Pearse RM. Mortality after surgery with SARS-CoV-2 infection in England: a population-wide epidemiological study. Br J Anaesth. 2021 Aug;127(2):205-214. doi: 10.1016/j.bja.2021.05.018. Epub 2021 Jun 11. PMID 34148733
- [Background] COVIDSurg Collaborative; GlobalSurg Collaborative. Timing of surgery following SARS-CoV-2 infection: an international prospective cohort study. Anaesthesia. 2021 Jun;76(6):748-758. doi: 10.1111/anae.15458. Epub 2021 Mar 9. PMID 33690889
- [Background] El-Boghdadly K, Cook TM, Goodacre T, Kua J, Denmark S, McNally S, Mercer N, Moonesinghe SR, Summerton DJ. Timing of elective surgery and risk assessment after SARS-CoV-2 infection: an update: A multidisciplinary consensus statement on behalf of the Association of Anaesthetists, Centre for Perioperative Care, Federation of Surgical Specialty Associations, Royal College of Anaesthetists, Royal College of Surgeons of England. Anaesthesia. 2022 May;77(5):580-587. doi: 10.1111/anae.15699. Epub 2022 Feb 22. PMID 35194788
- [Background] Mavrothalassitis O, Pirracchio R, Fong N, Lazzareschi D, Sharma A, Vaughn MT, Mathis M, Legrand M. Outcome of surgical patients during the first wave of the COVID-19 pandemic in US hospitals. Br J Anaesth. 2022 Jan;128(1):e35-e37. doi: 10.1016/j.bja.2021.09.023. Epub 2021 Oct 1. No abstract available. PMID 34689990
- [Background] Wijeysundera DN, Khadaroo RG. Surgery after a previous SARS-CoV-2 infection: data, answers and questions. Anaesthesia. 2021 Jun;76(6):731-735. doi: 10.1111/anae.15490. Epub 2021 Apr 17. No abstract available. PMID 33864692
- [Background] Lieberman N, Racine A, Nair S, Semczuk P, Azimaraghi O, Freda J, Eikermann M, Wongtangman K. Should asymptomatic patients testing positive for SARS-CoV-2 wait for elective surgical procedures? Br J Anaesth. 2022 May;128(5):e311-e314. doi: 10.1016/j.bja.2022.02.005. Epub 2022 Feb 16. No abstract available. PMID 35277245
- [Background] Dobbs TD, Gibson JAG, Fowler AJ, Abbott TE, Shahid T, Torabi F, Griffiths R, Lyons RA, Pearse RM, Whitaker IS. Surgical activity in England and Wales during the COVID-19 pandemic: a nationwide observational cohort study. Br J Anaesth. 2021 Aug;127(2):196-204. doi: 10.1016/j.bja.2021.05.001. Epub 2021 Jun 18. PMID 34148732
- [Derived] Zheng Z, Wang L, Wang S, Fan Q, Zhang H, Luo G, Gao B, Yang X, Zhao B, Wang X, Dong H, Nie H, Lei C. Inhaled Nitric Oxide ReDuce postoperatIve pulmoNAry complicaTions in patiEnts with recent COVID-19 infection (INORDINATE): protocol for a randomised controlled trial. BMJ Open. 2024 Mar 14;14(3):e077572. doi: 10.1136/bmjopen-2023-077572. PMID 38485487

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT05721144/SAP_000.pdf